Comparison of Clinpro™ 5000 1.1% Sodium Fluoride Anti-Cavity Toothpaste, Clinpro™ Tooth Crème, and MI-Paste Plus for the Prevention and Reduction of White Spot Lesions in Orthodontic Treatment

## **RESULTS AND STATISTICS**

The results will be evaluated in the following manner:

- (1) Difference in prevention of white spot formation between the control and the study groups using the EDI scores
- (2)Standard statistical methods were employed to analyze all data.

## DATA COLLECTION, DATABASE MANAGEMENT, AND DATA ANALYSIS

Data collection, database management, and data analyses were performed by sponsor personnel or its designee. Only the sponsor, or its appropriate designee, had access to individual-level patient data collected as part of this study, regardless of whether the patient provided informed consent and HIPAA authorization. All individual level patient data had identification information removed.



Figure 1. Enamel Decalcification Index. Facial surface of each tooth was divided into four areas. A score was allocated for each area of each tooth: 0=No decalcification to 3=Decalcifications covering 100% of the area.